CLINICAL TRIAL: NCT01908049
Title: Treatment With Probiotics (Saccharomyces Boulardii) and Its Role in Bacterial Translocation and Immune Reconstitution in VIH Infection.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, JVillar, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROB-VIH
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: HIV -1 Infection
Keywords: Probiotic; HIV; Microbial translocation; inflammation; microbiota composition
MeSH Terms: conditions — Inflammation | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): A probiotic (Saccharomyces boulardii) 2 caps/ 8h for 12 weeks.
  Interventions: Dietary Supplement: Probiotic.
- Placebo (Placebo Comparator): No active substance is given.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic.
  Arms: Probiotic
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Objectives: MAIN: To evaluate the parameters of microbial translocation after treatment with probiotics (Saccharomyces boulardii) in HIV+ patients and its role on immune reconstitution and the changes in gut microbiota composition.

SECONDARY OBJECTIVES: 1) To analyze the progress of immune activity markers after the administration of probiotics. 2) To determine the improvement of CD4+ lymphocytes and HIV viral load in patients after taking probiotics.

Methods: Design: A prospective randomized open controlled double-blinded trial, to be performed at a tertiary care hospital in Barcelona. Subjects: Chronic HIV infected patients. Sample size: 44 cases. They´ll be divided in 2 groups: (1) Patients with CD4 +> 400 cells / ml and undetectable viral load for more than two years (22 cases) and (2) Patients with immunodiscordancy, defined as patients with CD4 + T cells lower than 350 cells / ml despite 4-7 years of effective antiretroviral therapy. (22 cases). Intervention: Patients were randomized in 2 subgroups: (A) they´ll receive daily oral supplementation with S. boulardii for 3 months and (B) they ´ll receive placebo. Variables: bacterial lipopolisaccharide levels measured by the Lipid-Binding protein (LBP), parameters of immune activation in plasma (soluble CD14, IFN-Υ, TNF-Alpha, IL (interleukine)-2, IL-5, IL-6, IL-12)and gut microbiota composition prior to the use of probiotics (baseline), at 3 and 6 months. Immunological and clinical data. Outcome measures: quantification of bacterial translocation levels, markers of activity and immune recovery. Analysis: Comparison of variables before and after the intervention. The analysis will be performed by biological and immunological effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HIV infection and viral load undetectable > two years with stable ART CD4> 400 cells / ml.
* Patients with chronic HIV infection and viral load undetectable> two years with stable ART CD4 <350 cells / ml.
* Inform consent signed.
* Aged between 18- No limit.

Exclusion Criteria:

* Patients who receive or have received in the past 6 months food supplements containing probiotics.
* Patients who have received antibiotic treatment in the last two months
* Patients who are poor presupposes adherence to dietary supplements.
* Patients who have changed the TAR in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate microbial translocation-Binding lipopolysaccharide Protein (LBP). | From randomisation to 6 months.
To evaluate Gut microbiota composition. | From randomisation to 6 months.
  Change in gut microbiota (454 pyrosequencing of fecal samples).

SECONDARY OUTCOMES:
To evaluate Markers of immune activity: soluble CD14 (sCD14), interferon gamma (IFN-Υ), tumor necrosis factor (TNF), IL-6, Reactive C protein, D -dimer, fibrinogen. | From randomisation to 6 months.
Analyse parameters that determine the immune status: CD4 + lymphocyte count, CD 8 + and HIV viral load. | From randomisation to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Villar-Garcia J, Hernandez JJ, Guerri-Fernandez R, Gonzalez A, Lerma E, Guelar A, Saenz D, Sorli L, Montero M, Horcajada JP, Knobel Freud H. Effect of probiotics (Saccharomyces boulardii) on microbial translocation and inflammation in HIV-treated patients: a double-blind, randomized, placebo-controlled trial. J Acquir Immune Defic Syndr. 2015 Mar 1;68(3):256-63. doi: 10.1097/QAI.0000000000000468. PMID 25469528